CLINICAL TRIAL: NCT02736188
Title: Phase 3B Open-Label Extension Study to Evaluate the Safety and Efficacy of Aceneuramic Acid Extended-Release (Ace-ER) Tablets in Patients With GNE Myopathy (GNEM) or Hereditary Inclusion Body Myopathy (HIBM)
Brief Title: Study to Evaluate the Safety and Efficacy of Aceneuramic Acid Extended-Release (Ace-ER) Tablets in Patients With Glucosamine (UDP-N-acetyl)-2-epimerase Myopathy (GNEM) or Hereditary Inclusion Body Myopathy (HIBM)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX001-CL302
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hereditary Inclusion Body Myopathy; Distal Myopathy With Rimmed Vacuoles; Distal Myopathy, Nonaka Type; GNE Myopathy; Quadriceps Sparing Myopathy
Keywords: GNE Myopathy; GNEM; Nonaka; Hereditary Inclusion Body Myopathy; HIBM; DMRV; QSM
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: Aceneuramic Acid Extended-Release Tablets (Experimental): Participants will take 4 tablets (500 mg Ace-ER each for 2 g per dose) orally 3 times per day (TID).
  Interventions: Drug: Aceneuramic Acid Extended-Release Tablets

INTERVENTIONS:
Drug: Aceneuramic Acid Extended-Release Tablets
  Other Names: UX001; Sialic Acid Extended Release; Ace-ER

SUMMARY:
The objective of this study is to evaluate the long-term safety and efficacy of Ace-ER treatment in subjects with GNEM.

DETAILED DESCRIPTION:
This Phase 3b extension study will assess the long-term safety of Ace-ER in patients who participated in and completed study UX001-CL301 (NCT02377921), study UX001-CL202 (NCT01830972), and study UX001-CL203 (NCT02731690).

ELIGIBILITY:
Inclusion Criteria:

* Have completed UX001-CL202, UX001-CL301 or UX001-CL203 study
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and before any research-related procedures are conducted
* Willing to comply with all study procedures
* Female participants of child-bearing potential or male participants with female partners of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use a highly effective method of contraception as determined by the site investigator (i.e., oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation or true abstinence [when this is in line with the preferred and usual lifestyle of the subject], which means not having sex because the subject chooses not to), from the period following the signing of the informed consent through 30 days after last dose of study drug
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause for at least two years, have had tubal ligation at least one year prior to Screening, or who have had a total hysterectomy or bilateral salpingo oophorectomy

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

* Ingestion of N-acetyl-D-mannosamine (ManNAc) or related metabolites; intravenous immunoglobulin (IVIG); or anything that can be metabolized to produce SA in the body within 60 days prior to the Screening Visit
* Has had any hypersensitivity to sialic acid (SA) or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or anticipated requirement for any investigational agent prior to completion of all scheduled study assessments
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study
* Has a concurrent disease, active suicidal ideation, or other condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (14):
- United States (5):
  - UCLA, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Washington University School of Medicine, St. Louis, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
- UMHAT Alexandrovska, Bulgaria, Sofia, Bulgaria
- McMaster University, Hamilton, Ontario, Canada
- France (2):
  - CHU La Réunion - site GHSR, Saint-Pierre, Reunion
  - Institut de Myologie GH Pitié-Salpêtrière, Paris
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- Italy (3):
  - University of Messina, Messina
  - University of Milan, Milan
  - Università Cattolica, Rome
- The Newcastle upon Tyne Hospitals, Newcastle upon Tyne, Tyne and Wear, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 143 participants were screened and enrolled across 14 total sites in the United States, Israel, United Kingdom, Italy, France, Canada, and Bulgaria. 87 participants rolled over from study UX001-CL301 (NCT02377921), 49 participants rolled over from study UX001-CL202 (NCT01830972), and 7 participants rolled over from UX001-CL203 (NCT02731690).
Pre-assignment Details: Of the143 participants who enrolled, 1 participant withdrew consent prior to receiving the first dose and is not included in the Safety Analysis Population presented below.
Groups:
- Ace-ER 6 g/Day: 4 tablets (500 mg Ace-ER each for 2 g per dose) orally 3 times per day
Period: Overall Study
Arm/Group | Ace-ER 6 g/Day
Started | 142
Completed | 0
Not Completed | 142
Not completed — Discontinuation of Study by Sponsor | 134
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least one dose of study drug in UX001-CL302.
Arm/Group | Ace-ER 6 g/Day
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 125
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 111
  Asian | 19
  Other, Not Specified | 12
Hand Held Dynamometry (HHD) Upper Extremity Composite Score (UEC) [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kilogram-force [kgf]) for each was recorded. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  kgf
    number analyzed (Participants) | 87
    (all) | 52.98 (28.814)
Glucosamine (UDP-N-acetyl)-2-epimerase Myopathy Functional Activities Scale(GNEM-FAS) Mobility Score [Mean (Standard Deviation); unit: score on a scale] — GNEM-FAS Expanded Version Mobility subscale score has 13 items and ranges from 0 to 52 with higher scores representing greater mobility. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  score on a scale
    number analyzed (Participants) | 87
    (all) | 24.17 (7.772)
GNEM-FAS Expanded Version Upper Extremity Score [Mean (Standard Deviation); unit: score on a scale] — GNEM-FAS Expanded Version Upper Extremity subscale score has 9 items and ranges from 0 to 36 with higher scores representing more skilled, independent use of the arms during functional activity performance. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  score on a scale
    number analyzed (Participants) | 87
    (all) | 27.53 (4.938)
HHD Lower Extremity Composite (LEC) Score [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  kgf
    number analyzed (Participants) | 86
    (all) | 51.91 (37.474)
Sit-to-Stand Test [Mean (Standard Deviation); unit: stands] — Lower extremity function was assessed using a sit-to-stand test. The number of times the participant can rise from a seated to a standing position in a 30-second period was recorded. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  stands
    number analyzed (Participants) | 87
    (all) | 12.75 (4.977)
30-second Weighted Arm Lift Test [Mean (Standard Deviation); unit: lifts] — Upper extremity function was assessed using a weighted arm lift test performed bilaterally. The number of times the participant can raise a 1 kg weight above the head in a 30-second period was recorded. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  lifts
    number analyzed (Participants) | 72
    (all) | 30.93 (13.171)
Six-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — The total distance walked (meters) in a 6-minute period was measured. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  meters
    number analyzed (Participants) | 83
    (all) | 359.4 (123.94)
Percent Predicted Meters Walked in 6MWT [Mean (Standard Deviation); unit: percentage of predicted meters] — The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated. Predicted 6MWT distance (meters) = 868.8 - (2.99 x Age) - (74.7 x Sex), where age is baseline age in years, and sex = 0 for males, and 1 for females. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  percentage of predicted meters
    number analyzed (Participants) | 83
    (all) | 49.52 (16.962)
Total Force in Knee Extensors [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  kgf
    number analyzed (Participants) | 84
    (all) | 26.60 (9.746)
Percent of Predicted Total Force in Knee Extensors [Mean (Standard Deviation); unit: percent of predicted total force] — The percent predicted total force value of lower extremity muscle strength in the knee extensors was determined based on reference equations adjusting for age, gender, height, and weight. Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
  percent of predicted total force
    number analyzed (Participants) | 81
    (all) | 13.69 (15.323)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious AEs (SAEs), and Discontinuations Due to AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug, whether or not considered drug related. An SAE or serious suspected adverse reaction is an AE or suspected adverse reaction that at any dose, in the view of either the Investigator or Ultragenyx, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect. TEAEs were defined as any AE that occurred after the first dose of study drug. The severity of all AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03: grade1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening, grade 5=death.
Time Frame: From first dose of study drug through the end of treatment plus 30 days (+5 days). Mean (SD) duration of treatment was 256.3 (101.54) days.
Population: Safety Analysis Set: all participants who received at least one dose of study drug in UX001-CL302.
Measure: Count of Participants; unit: Participants
Arm/Group | Ace-ER 6 g/Day
Number analyzed (Participants) | 142
Participants
  TEAEs | 104
  Serious TEAEs (SAEs) | 7
  Deaths | 0
  Grade 3 or 4 TEAEs | 11
  TEAEs Leading to Study Drug Discontinuation | 2
  TEAEs Leading to Study Discontinuation | 1

2. Primary Outcome: Change From Baseline in HHD UEC Score Over Time
Description: Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. The UEC is derived from the sum of the average of the right and left total force (measured in kgf). Analyzed using a repeated measure generalized estimation equation (GEE) model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, 48
Population: Full Analysis Set: all participants in parent study UX001-CL301 (NCT02377921) with a UX001-CL302 baseline measurement and at least one post-baseline measurement in UX001-CL302.
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Groups:
- Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day): 4 tablets (500 mg Ace-ER each for 2 g per dose) orally 3 times per day in participants who took Ace-ER in study UX001-CL301 (NCT02377921)
- Ace-ER 6 g/Day (Parent Study Treatment: Placebo): 4 tablets (500 mg Ace-ER each for 2 g per dose) orally 3 times per day in participants who took placebo in study UX001-CL301 (NCT02377921)
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
kgf
  Week 8 | 0.88 [-0.75 to 2.51] | 0.09 [-1.05 to 1.23]
  Week 16 | 0.10 [-1.47 to 1.67] | -0.26 [-1.26 to 0.74]
  Week 24 | -1.40 [-2.92 to 0.12] | -0.49 [-2.13 to 1.15]
  Week 48 | -2.24 [-4.95 to 0.47] | -2.18 [-4.30 to -0.07]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.4287, generalized estimating equation (GEE) — Baseline is fit into the model as a covariate; LS Mean Difference = 0.80, 95% CI 2-sided [-1.17 to 2.77]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.7031, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = 0.36, 95% CI 2-sided [-1.49 to 2.21]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.4253, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = -0.91, 95% CI 2-sided [-3.14 to 1.32]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.9747, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = -0.06, 95% CI 2-sided [-3.49 to 3.38]

3. Secondary Outcome: Change From Baseline in the GNEM-FAS Expanded Version Mobility Domain Score Over Time
Description: GNEM-FAS Expanded Version Mobility subscale score has 13 items and ranges from 0 to 52 with higher scores representing greater mobility. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
score on a scale
  Week 8 | -0.12 [-0.66 to 0.42] | 0.15 [-0.35 to 0.65]
  Week 16 | -0.30 [-0.87 to 0.27] | -0.12 [-0.72 to 0.49]
  Week 24 | -0.78 [-1.31 to -0.25] | -0.34 [-0.92 to 0.23]
  Week 48 | -0.73 [-1.43 to -0.03] | -0.45 [-1.67 to 0.77]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.4721, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = -0.27, 95% CI 2-sided [-1.01 to 0.47]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.6611, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = -0.19, 95% CI 2-sided [-1.02 to 0.64]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.2760, GEE model; Baseline is fit into the model as a covariate; LS Mean Difference = -0.44, 95% CI 2-sided [-1.22 to 0.35]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.6977, GEE model — Baseline is fit into the model as a covariate; LS Mean Difference = -0.28, 95% CI 2-sided [-1.69 to 1.13]

4. Secondary Outcome: Change From Baseline on the GNEM-FAS Upper Extremity Domain Score Over Time
Description: GNEM-FAS Expanded Version Upper Extremity subscale score has 9 items and ranges from 0 to 36 with higher scores representing more skilled, independent use of the arms during functional activity performance. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
score on a scale
  Week 8 | 0.68 [0.15 to 1.22] | -0.02 [-0.55 to 0.51]
  Week 16 | 0.34 [-0.21 to 0.89] | -0.40 [-0.99 to 0.19]
  Week 24 | 0.26 [-0.41 to 0.93] | -0.17 [-1.01 to 0.67]
  Week 48 | -0.82 [-2.16 to 0.51] | -0.48 [-1.03 to 0.07]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.0648, GEE model — Baseline is fit into the model as a covariate; Difference in LS Means = 0.70, 95% CI 2-sided [-0.04 to 1.45]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.0692, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.74, 95% CI 2-sided [-0.06 to 1.55]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.4317, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.44, 95% CI 2-sided [-0.65 to 1.52]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.6416, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.34, 95% CI 2-sided [-1.78 to 1.10]

5. Secondary Outcome: Change From Baseline in HHD Lower Extremity Composite (LEC) Score Over Time
Description: Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. The LEC is derived from the sum of the average of the right and left total force (measured in kgf). Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
kgf
  Week 8 | 0.01 [-2.01 to 2.04] | -0.77 [-3.65 to 2.11]
  Week 16 | -1.63 [-3.95 to 0.34] | -0.98 [-3.77 to 1.81]
  Week 24 | -0.60 [-3.90 to 2.71] | -0.10 [-3.82 to 3.62]
  Week 48 | -0.32 [-4.02 to 3.39] | -4.47 [-7.45 to -1.49]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.6546, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.78, 95% CI 2-sided [-2.65 to 4.22]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.7054, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.64, 95% CI 2-sided [-3.97 to 2.69]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.8441, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.50, 95% CI 2-sided [-5.45 to 4.45]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.0864, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 4.15, 95% CI 2-sided [-0.59 to 8.90]

6. Secondary Outcome: Change From Baseline in the Number of Stands in the Sit-to-Stand Test Over Time
Description: Lower extremity function was assessed using a sit-to-stand test. The number of times the participant can rise from a seated to a standing position in a 30-second period was recorded. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: stands
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
stands
  Week 8 | 0.02 [-0.43 to 0.46] | -0.05 [-0.61 to 0.51]
  Week 16 | -0.04 [-0.49 to 0.40] | 0.14 [-0.39 to 0.66]
  Week 24 | 0.06 [-0.43 to 0.56] | -0.41 [-0.94 to 0.12]
  Week 48 | -0.39 [-1.36 to 0.57] | -0.36 [-1.11 to 0.39]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.8603, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.06, 95% CI 2-sided [-0.65 to 0.78]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.6154, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.18, 95% CI 2-sided [-0.86 to 0.51]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.1999, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.47, 95% CI 2-sided [-0.25 to 1.20]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.9568, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.03, 95% CI 2-sided [-1.25 to 1.18]

7. Secondary Outcome: Change From Baseline in Number of Lifts in the 30-Second Weighted Arm Lift Test Over Time
Description: Upper extremity function was assessed using a weighted arm lift test performed bilaterally. The number of times the participant can raise a 1 kg weight above the head in a 30-second period was recorded. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: lifts
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
lifts
  Week 8 | 0.26 [-1.00 to 1.52] | -0.19 [-0.90 to 0.53]
  Week 16 | 0.03 [-1.22 to 1.27] | 0.59 [-0.50 to 1.68]
  Week 24 | 0.13 [-0.98 to 1.24] | -0.14 [-1.33 to 1.06]
  Week 48 | -1.58 [-3.60 to 0.45] | -1.17 [-2.55 to 0.22]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.5447, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.45, 95% CI 2-sided [-1.00 to 1.90]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.5051, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.56, 95% CI 2-sided [-2.22 to 1.09]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.7478, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.27, 95% CI 2-sided [-1.36 to 1.90]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.7429, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.41, 95% CI 2-sided [-2.86 to 2.04]

8. Secondary Outcome: Change From Baseline in Meters Walked in 6MWT Over Time
Description: The total distance walked (meters) in a 6-minute period was measured. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
meters
  Week 8 | -1.40 [-8.34 to 5.53] | -3.41 [-7.92 to 1.10]
  Week 16 | -3.91 [-12.03 to 4.20] | -1.93 [-8.32 to 4.47]
  Week 24 | -2.73 [-10.81 to 5.35] | -6.88 [-13.43 to -0.33]
  Week 48 | -13.91 [-25.58 to -2.25] | -21.89 [-38.51 to -5.28]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.6434, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 2.00, 95% CI 2-sided [-6.48 to 10.49]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.7118, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -1.99, 95% CI 2-sided [-12.53 to 8.55]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.4399, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 4.15, 95% CI 2-sided [-6.39 to 14.69]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.4430, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 7.98, 95% CI 2-sided [-12.41 to 28.37]

9. Secondary Outcome: Change From Baseline in Percent Predicted Meters Walked in 6MWT Over Time
Description: The total distance walked (meters) in a 6-minute period was measured, and the percent predicted distance based on normative data for age and gender was estimated. Predicted 6MWT distance (meters) = 868.8 - (2.99 x Age) - (74.7 x Sex), where age is baseline age in years, and sex = 0 for males, and 1 for females. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of predicted distance
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
percent of predicted distance
  Week 8 | -0.17 [-1.12 to 0.79] | -0.45 [-1.09 to 0.20]
  Week 16 | -0.49 [-1.60 to 0.61] | -0.24 [-1.15 to 0.67]
  Week 24 | -0.38 [-1.49 to 0.73] | -0.96 [-1.88 to -0.03]
  Week 48 | -1.94 [-3.56 to -0.31] | -2.93 [-5.04 to -0.81]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.6428, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.28, 95% CI 2-sided [-0.90 to 1.46]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.7334, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.25, 95% CI 2-sided [-1.72 to 1.21]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.4409, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.58, 95% CI 2-sided [-0.89 to 2.04]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.4687, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.99, 95% CI 2-sided [-1.69 to 3.68]

10. Secondary Outcome: Change From Baseline in Total Force in Knee Extensors Over Time
Description: Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Bilateral total force was defined as the average of the right and left force (measured in kgf). Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
kgf
  Week 8 | 0.50 [-0.77 to 1.78] | -0.64 [-1.53 to 0.25]
  Week 16 | -0.95 [-2.03 to 0.14] | -0.75 [-2.05 to 0.55]
  Week 24 | 0.33 [-1.33 to 2.00] | -0.46 [-2.15 to 1.23]
  Week 48 | 0.63 [-2.30 to 3.56] | -0.08 [-2.28 to 2.13]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.1502, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 1.14, 95% CI 2-sided [-0.41 to 2.69]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.8188, GEE model — Baseline is fit into the model as a covariate; difference in LS means = -0.20, -1.89% CI 2-sided [-1.89 to 1.49]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.5122, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.80, 95% CI 2-sided [-1.58 to 3.17]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.7022, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.72, 95% CI 2-sided [-2.96 to 4.40]

11. Secondary Outcome: Change From Baseline in Percent Predicted Total Force in Knee Extensors Over Time
Description: The percent predicted total force value of lower extremity muscle strength in the knee extensors was determined based on reference equations adjusting for age, gender, height, and weight. Analyzed using a repeated measure GEE model, which includes the baseline value as a covariate.
Time Frame: Baseline, Weeks 8, 16, 24, and 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of predicted total force (kgf)
Arm/Group | Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) | Ace-ER 6 g/Day (Parent Study Treatment: Placebo)
Number analyzed (Participants) | 44 | 43
percent of predicted total force (kgf)
  Week 8 | -0.98 [-1.78 to -0.19] | -1.17 [-2.44 to 0.09]
  Week 16 | -0.59 [-1.48 to 0.31] | -1.25 [-2.43 to -0.07]
  Week 24 | -0.70 [-1.92 to 0.53] | -0.85 [-2.53 to 0.83]
  Week 48 | -1.02 [-2.17 to 0.13] | -3.10 [-4.40 to -1.80]
Statistical Analysis 1: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 8; Test type: Superiority; p = 0.7906, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.19, 95% CI 2-sided [-1.22 to 1.60]
Statistical Analysis 2: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 16; Test type: Superiority; p = 0.3531, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.66, 95% CI 2-sided [-0.74 to 2.07]
Statistical Analysis 3: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 24; Test type: Superiority; p = 0.8846, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 0.15, 95% CI 2-sided [-1.92 to 2.23]
Statistical Analysis 4: Comparison: Ace-ER 6 g/Day (Parent Study Treatment: Ace-ER 6 g/Day) vs Ace-ER 6 g/Day (Parent Study Treatment: Placebo); Week 48; Test type: Superiority; p = 0.0168, GEE model — Baseline is fit into the model as a covariate; difference in LS means = 2.08, 95% CI 2-sided [0.38 to 3.79]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment plus 30 days (+5 days). Mean (SD) duration of treatment was 256.3 (101.54) days.
Arm/Group | Ace-ER 6 g/Day
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 7/142
Other Adverse Events (participants affected / at risk) | 66/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=142)
Abdominal pain (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Atypical pneumonia (Infections and infestations) | 1
Biopsy kidney (Investigations) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal pain (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=142)
Diarrhoea (Gastrointestinal disorders) | 10
Flatulence (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 8
Fall (Injury, poisoning and procedural complications) | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 17
Back pain (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 8

LIMITATIONS AND CAVEATS:
No efficacy result summaries or analyses were performed for participants rolling over from UX001-CL202 or UX001-CL203 because of the limited data from those participants due to the early study closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT02736188/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02736188/SAP_000.pdf